CLINICAL TRIAL: NCT04328428
Title: The Evaluation of Single Acupoint Therapy to Acute Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202000002A3
Record Dates: First submitted 2020-03-29; First posted 2020-03-31 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-02

CONDITIONS: Acupuncture; Acute Low Back Pain
Keywords: acute low back pain; BL40; Extra Meridian 32 (EM32); acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: three groups randomly:experiment group and two control groups. Patients in experiment group receive modified BL40 acupuncture. Control group one receives EM32 acupuncture and control group two receives BL40 acupuncture
Who Masked: Participant
Masking Description: The participants only know that they accept acupuncture ,but do not know which acupoint needling they receive.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (A)modified BL40 acupuncture (Experimental): modified BL40 acupuncture Participants receive BL40 acupuncture once on the same site of low back pain.
  Interventions: Other: acupuncture
- (B)EM32 acupuncture (Active Comparator): EM32 acupuncture Participants receive EM32 acupuncture once on the opposite site.
  Interventions: Other: acupuncture
- (C)BL40 acupuncture (Active Comparator): BL40 acupuncture Participants receive BL40 acupuncture once on the same site of low back pain
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Use one acupuncture needle insert in a acupoint.

SUMMARY:
Low back pain is the leading course of disability , affecting patients' health and work.

Recently, studies have reveal the fact that patients get insufficient physical activity and easily let acute stage turn to chronic type.

Although acupuncture for low back pain is worldwide popular, the mechanism of single acupoint for low back pain is still unclear.

Therefore, the aim of this study is the investigators choose the most frequent used acupoint and modified single acupoint method to assess the efficacy of single acupoint to acute low back pain.

DETAILED DESCRIPTION:
Low back pain is the leading course of disability , affecting patients' health and work. According to the study in 2013, 8.9 percent people of the world experienced over three months low back pain.

Recently, studies have reveal the fact that patients get insufficient physical activity and easily let acute stage turn to chronic type.

Although acupuncture for low back pain is worldwide popular, the mechanism of single acupoint for low back pian is still unclear.

Therefore, the investigators choose the most frequent used acupoint and modified single acupoint method to assess the efficacy of single acupoint to acute low back pain.

The investigators would like to compare the efficacy of the modified Bladder 40 (BL40) acupuncture to single acupoint through statistical analysis.

The investigators expect that all group will alleviate low back pain. However, treatment group will have statistical difference compared with control groups.

The aim of this study is the investigators choose the most frequent used acupoint and modified single acupoint method to assess the efficacy of single acupoint to acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* low back pain,duration < 1 month
* accept subject consent

Exclusion Criteria:

* without X ray or MRI image
* severe trauma , fracture or spondylosis found from image ,progression neurological symptoms suspected from central nerve system, rheumatic disease, fever or infection is suspected ,weight or cancer history , pregnancy and psychiatric disorder or not able to communication .

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-28 (Estimated); Primary Completion 2021-02-12 (Estimated); Study Completion 2021-02-12 (Estimated)

PRIMARY OUTCOMES:
pain measurement | 30 minutes
  use Visual Analogue Scale to measure pain intensity and algometer to measure pain threshold The minimum of Visual Analogue Scale is 0 and maximum values is 10. The higher Visual Analogue Scale mean a worse outcome . Newton is used to measure pain threshold. The higher pain threshold scores mean a better outcome .
range of motion measurement | 30 minutes
  measure the range of motion when lumbar extension and flexion

CONTACTS AND LOCATIONS:
Overall Officials: Ko-Hung Lee, MD, Study Chair — ChangGung Memorial Hospital
Locations (1):
- Dept of Chinese medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Hong J, Reed C, Novick D, Happich M. Costs associated with treatment of chronic low back pain: an analysis of the UK General Practice Research Database. Spine (Phila Pa 1976). 2013 Jan 1;38(1):75-82. doi: 10.1097/BRS.0b013e318276450f. PMID 23038621
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Asmundson GJG, Norton RG, Allerdings MD. Fear and avoidance in dysfunctional chronic back pain patients. Pain. 1997 Feb;69(3):231-236. doi: 10.1016/S0304-3959(96)03288-5. PMID 9085296
- [Background] Kent PM, Keating JL. Can we predict poor recovery from recent-onset nonspecific low back pain? A systematic review. Man Ther. 2008 Feb;13(1):12-28. doi: 10.1016/j.math.2007.05.009. Epub 2007 Jul 19. PMID 17658288
- [Background] Vas J, Aranda JM, Modesto M, Benitez-Parejo N, Herrera A, Martinez-Barquin DM, Aguilar I, Sanchez-Araujo M, Rivas-Ruiz F. Acupuncture in patients with acute low back pain: a multicentre randomised controlled clinical trial. Pain. 2012 Sep;153(9):1883-1889. doi: 10.1016/j.pain.2012.05.033. Epub 2012 Jul 4. PMID 22770838